CLINICAL TRIAL: NCT02727894
Title: Colorectal Cancer Screening Detects Tumors at Earlier Stages Improving Clinical Outcomes
Brief Title: Colorectal Cancer: Screening vs. Non-Screening
Acronym: CRC
Status: Completed | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Private practice at Hluboká nad Vltavou (Unknown); Klaudian Hospital Mladá Boleslav (Unknown); Masaryk Hospital Usti nad Labem (Other); Brno University Hospital (Other); Medic Kral Ltd. (Unknown); Chomutov Hospital (Unknown); Tomas Bata Hospital, Czech Republic (Other); Military University Hospital, Prague (Other); Frýdek-Místek Hospital (Unknown); The University Hospital Plzeň (Unknown); Vitkovice Hospital (Other)
Responsible Party: Principal Investigator, Jan Král, MD, M.D., Institute for Clinical and Experimental Medicine
Other Study IDs: 00023001-2015
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer; Screening
Keywords: Screening; pTNM; Metastasis; Chemotherapy; Resection Margins; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Margins of Excision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Screening Group: CRC diagnosed by screening was defined as cancer diagnosed by primary screening colonoscopy, or colonoscopy after a positive immunochemical based faecal occult blood test i(FOBT) in patients without symptoms invited to examination according to the national screening programme policy
- Non-screening Group: Symptomatic CRC was defined as cancer diagnosed in symptomatic patients.

SUMMARY:
The purpose of this study is to determine whether colorectal cancer diagnosed by screening (primary screening colonoscopy, colonoscopy after immunochemical based faecal occult blood test) has more favourable clinical-pathological characteristics than colorectal cancer diagnosed for symptoms. We aimed to compare these two groups of patients at the time of diagnosis and confirm the efficiency of the screening programme.

DETAILED DESCRIPTION:
Multicentre prospective observational study. 12 centres across the Czech rep. included. Study approved by Ethical Committee.

All participants gave their informed signed consent. Each centre was assigned a unique ID number to distinguish between the locations in which patients were enrolled.

Patients informations were stored under identification number in secure internet database (RedCap) run by The International Clinical Research Center of St. Anne's University Hospital Brno.REDCap is a secure, web-based application designed to support data capture for research studies.

Statistical analysis was done with SAS, ver. 9.3. Descriptive statistics such as absolute and relative frequencies and median with 95 % confidence intervals were used. Differences between the screening and non-screening groups were compared using the Chi-square test or Fisher's exact test (categorical parameters) and Mann-Whitney test (continuous parameters). Results with a p-value < 0.05 were considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed colorectal cancer

Exclusion Criteria:

* unsigned informed consent
* mental disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinics, university hospitals, private practices
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Král, M.D., Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 2013 till September 2015 in 12 centres across the Czech Republic 276 patients were enrolled.
Pre-assignment Details: Patients with diagnosed colorectal carcinoma were enrolled (276). 11 patients were excluded because of the inability to categorise those patients into the screening or non-screening group.
Groups:
- Screening Group: CRC diagnosed by screening was defined as cancer diagnosed by primary screening colonoscopy, or colonoscopy after a positive immunochemical based faecal occult blood test (iFOBT) in patients without symptoms invited to examination according to the national screening programme policy
Period: Overall Study
Arm/Group | Screening Group | Non-screening Group
Started | 73 (March 2013) | 192 (March 2013)
Completed | 73 (September 2015) | 192 (September 2015)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Screening: Patients with colorectal cancer diagnosed by screening procedures (primary screening colonoscopy, colonoscopy after FOBT).
- Others: Patients with colorectal cancer diagnosed by other diagnostic procedures (diagnostic colonoscopy, CT, magnetic resonance, ultrasonography, urgent surgery, etc.)
- Total: Total of all reporting groups
Arm/Group | Screening | Others | Total
Number analyzed (Participants) | 73 | 192 | 265
Age, Customized [Median (Full Range); unit: years]
  Age (years, median) | 67.5 [39 to 91] | 70 [33 to 91] | 68 [33 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 77 | 106
  Male | 44 | 115 | 159

OUTCOME MEASURES:

1. Primary Outcome: Colorectal Cancer Stage (pTNM)
Description: Differences between colorectal cancer stage (0,I,II) in screening vs. non-screening group.
  * 0. stage (Tis N0 M0)
  * I. stage (T1-2 N0 M0)
  * II. stage (T3-4 N0 M0)
  * III. stage (T1-4 N1-2 M0)
  * IV. stage (T1-4 N1-2 M1)
  Stages 0,I II were considered to have better outcome
Time Frame: at time of diagnosis
Measure: Count of Participants; unit: Participants
Groups:
- Screening Group: Patients with colorectal cancer diagnosed by screening procedures (primary screening colonoscopy, colonoscopy after iFOBT).
- Non-Screening Group: Symptomatic CRC was defined as cancer diagnosed in symptomatic patients by colonoscopy, or by CT, MRI or ultrasonography before verification by colonoscopy.
Arm/Group | Screening Group | Non-Screening Group
Number analyzed (Participants) | 73 | 192
Participants | 46 | 85

2. Secondary Outcome: Colorectal Cancer Grade
Description: Differences between colorectal cancer grade in screening vs. non-screening group.
  * GX (cannot be identified)
  * G1 (well diff.)
  * G2 (moderately diff.)
  * G3 (poorly diff.)
  * G4 (undifferentiated)
  Grades 1,2 were considered to have connection with lower stage
Time Frame: after surgery was performed
Measure: Count of Participants; unit: Participants
Groups:
- Screening Group: Patients with colorectal cancer diagnosed by screening (primary screening colonoscopy, colonoscopy after iFOBT).
- Non-screening Group: Symptomatic CRC (non-screening group) was defined as cancer diagnosed in symptomatic patients by colonoscopy, or by CT, MRI or ultrasonography before verification by colonoscopy.
Arm/Group | Screening Group | Non-screening Group
Number analyzed (Participants) | 73 | 192
Participants | 53 | 120

3. Secondary Outcome: Colorectal Cancer Resection Margins
Description: Difference between colorectal cancer resection margins (RX, R0, R1, R2) in screening vs. non-screening group.
  * RX: cannot be identified
  * R0: no cancer cells seen microscopically at the resection margin
  * R1: cancer cells present microscopically at the resection margin (microscopic positive margin)
  * R2: gross examination by the naked eye shows tumor tissue present at the resection margin (macroscopic positive margin)
Time Frame: after surgery was performed
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Group | Non-screening Group
Number analyzed (Participants) | 62 | 154
Participants | 48 | 94

4. Secondary Outcome: Colorectal Cancer Metastasis
Description: Differences between occurrence of colorectal cancer metastasis (MX, M0, M1) between screening vs. non-screening group.
  * MX: cannot be measured
  * M0: cancer has not spread to other parts of the body
  * M1: cancer has spread to other parts of the body
Time Frame: at time of diagnosis
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Group | Non-Screening Group
Number analyzed (Participants) | 73 | 192
Participants | 55 | 104

5. Secondary Outcome: Colorectal Cancer Surgery
Description: Median time between diagnosis and surgery.
Time Frame: time between diagnosis and surgery, measured after surgery was performed
Measure: Median (95% Confidence Interval); unit: Number of day betw. diagnosis and surg.
Arm/Group | Screening Group | Non-Screening Group
Number analyzed (Participants) | 73 | 192
Number of day betw. diagnosis and surg. | 30 [24 to 35] | 21.5 [19 to 24]

6. Secondary Outcome: Colorectal Cancer and Palliative Therapy
Description: Differences between neoadjuvant, adjuvant and systemic palliative therapy in screening vs. non-screening group.
  Number of patients treated with palliative therapy in both groups.
Time Frame: during treatment plan setting
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Group | Non-Screening Group
Number analyzed (Participants) | 73 | 192
Participants | 2 | 23

ADVERSE EVENTS:
Description: Adverse event data were not collected because data were mainly obtained at the time of diagnosis or at the time of treatment plan setting.
  Study was focused on comparing screening group and non-screening group at the time of diagnosis and confirm the efficiency of the screening programme.
Groups:
- Screening Group: Patients with colorectal cancer diagnosed by screening (primary screening colonoscopy, colonoscopy after FOBT).
- Non-screening Group: Symptomatic CRC was defined as carcinoma detected by CT, MR or sonography and then verified by colonoscopy.
Arm/Group | Screening Group | Non-screening Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results can be published exclusively by the main investigator or after main investigator approval.